CLINICAL TRIAL: NCT05752461
Title: A Multicenter, Randomized, Active-comparator-controlled Phase 2 Clinical Trial to Assess the Efficacy and Safety of a Single Subcutaneous Injection of SHR-2004 in Patients Undergoing Elective Unilateral Total Knee Arthroplasty
Brief Title: SHR-2004 for the Prevention of Venous Thromboembolism in Patients Undergoing Total Knee Arthroplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Suncadia Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SHR-2004-201
Record Dates: First submitted 2023-02-22; First posted 2023-03-02 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Prevention of Venous Thromboembolism After Knee Arthroplasty
MeSH Terms: interventions — enoxaparin sodium

STUDY DESIGN:
Intervention Model Description: SHR-2004 injection compared with Enoxaparin sodium injection
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment group A: SHR-2004 injection (Experimental)
  Interventions: Drug: SHR-2004 injection
- Treatment group B: SHR-2004 injection (Experimental)
  Interventions: Drug: SHR-2004 injection
- Treatment group C: SHR-2004 injection (Experimental)
  Interventions: Drug: SHR-2004 injection
- Treatment group D: Enoxaparin sodium injection (Active Comparator)
  Interventions: Drug: Enoxaparin sodium injection

INTERVENTIONS:
Drug: SHR-2004 injection — low dose subcutaneous injection once
  Arms: Treatment group A: SHR-2004 injection
Drug: SHR-2004 injection — medium dose subcutaneous injection once
  Arms: Treatment group B: SHR-2004 injection
Drug: SHR-2004 injection — high dose subcutaneous injection once
  Arms: Treatment group C: SHR-2004 injection
Drug: Enoxaparin sodium injection — 40 mg administered as subcutaneous injection once daily
  Arms: Treatment group D: Enoxaparin sodium injection

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of SHR-2004 in preventing venous thromboembolism after elective unilateral total knee arthroplasty

ELIGIBILITY:
Inclusion Criteria:

1. Understand the research procedures and methods, volunteer to participate in the study, and sign the informed consent
2. Scheduled to undergo elective unilateral total knee arthroplayts (TKA)
3. Male or female(≥ 40 years old and < 80 years old)

Exclusion Criteria:

1. Unable to receive CT angiography of both lower limbs;
2. Malignant tumor within one year of the screening ;
3. History of venous thromboembolism;
4. Myocardial infarction, transient ischemic attack or ischemic stroke occurred within 6 months of the screening;
5. Any medical history that may increase the risk of bleeding or any conditions that the investigator considers to increase the risk of bleeding
6. Any of the laboratory test indicators meets the following criteria:

   ①estimated Glomerular Filtration Rate < 60 mL/min/1.73m2 ;

   ②Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 times the upper limit of normal value (ULN);

   ③total bilirubin was > 2 times, etc
7. History of drug abuse;
8. Pregnant or lactating women

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Incidence of composite endpoint consisting of asymptomatic DVT as detected by mandatory bilateral CT venography, confirmed symptomatic DVT, non-fatal PE and all-cause death（Primary efficacy outcome） | Day 12
Incidence of composite endpoint of major and clinically relevant non-major bleeding（Primary safety outcome） | Day 12

SECONDARY OUTCOMES:
Incidence of composite endpoint consisting of asymptomatic DVT as detected by mandatory bilateral CT venography, confirmed symptomatic DVT, non-fatal PE and all-cause death（Secondary efficacy endpoint） | Day 85
Incidence of composite endpoint of any bleeding（Secondary safety endpoint） | Day 12
Incidence of composite endpoint of major and clinically relevant non-major bleeding（Secondary safety endpoint） | Day 85

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided